CLINICAL TRIAL: NCT04560673
Title: Optimizing Neurofeedback to Treat Chemotherapy Induced Peripheral Neuropathy
Brief Title: Duloxetine and Neurofeedback Training for the Treatment of Chemotherapy Induced Peripheral Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0712; NCI-2020-06553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0712 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Duloxetine Hydrochloride; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (neurofeedback training, duloxetine) (Experimental): Patients receive neurofeedback training over 1 hour 3-5 times weekly for up to 5 weeks. Patients also receive duloxetine PO QD for 5 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: Duloxetine; Behavioral: Neurofeedback; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (neurofeedback training) (Experimental): Patients receive neurofeedback training over 1 hour 3-5 times weekly for up to 5 weeks.
  Interventions: Behavioral: Neurofeedback; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (duloxetine) (Experimental): Patients receive duloxetine PO QD for 5 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: Duloxetine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Duloxetine — Given PO
  Arms: Group I (neurofeedback training, duloxetine); Group III (duloxetine)
Behavioral: Neurofeedback — Receive neurofeedback training
  Other Names: EEG biofeedback
  Arms: Group I (neurofeedback training, duloxetine); Group II (neurofeedback training)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial investigates how well duloxetine and neurofeedback training work in treating patients with chemotherapy induced peripheral neuropathy. Duloxetine is a type of serotonin and norepinephrine reuptake inhibitor that increases the amount of certain chemicals in the brain that help relieve depression and peripheral neuropathy. Neurofeedback training is a type of therapy that uses an electroencephalograph (EEG) and a computer software program to measure brain wave activity and may help teach patients with peripheral neuropathy (nerve damage) how to change their own brain waves to lower their feelings of neuropathy and help improve their overall quality of life. Giving duloxetine and neurofeedback training may work better in treating peripheral neuropathy caused by chemotherapy compared to duloxetine or neurofeedback training alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine if the combination of duloxetine (DL) and neurofeedback (NFB) is superior to DL or NFB alone in treating chemotherapy induced peripheral neuropathy (CIPN).

SECONDARY OBJECTIVES:

I. Determine the optimal number of neurofeedback sessions needed to result in long-term relief of CIPN in a large cohort of cancer survivors and across socioeconomic groups.

II. Examine baseline brain signatures as a predictor of response to neurofeedback (NFB) and to duloxetine and determine who will require more sessions of NFB to achieve relief of symptoms.

III. Examine if the combination of DL + NFB (than those getting DL or NFB alone) or a larger number of NFB sessions results in better improvements in cancer-related symptoms, physical functioning, and quality of life (QOL).

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients receive neurofeedback training over 1 hour each 3-5 times weekly for up to 5 weeks. Patients also receive duloxetine orally (PO) once daily (QD) for 5 weeks in the absence of unacceptable toxicity.

GROUP II: Patients receive neurofeedback training session over 1 hour 3-5 times weekly for up to 5 weeks.

GROUP III: Patients receive duloxetine PO QD for 5 weeks in the absence of unacceptable toxicity.

After completion of study, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Pain score >= 4 on a 0-10 numeric pain scale and/or grade 1-4 neuropathic pain according to the National Cancer Institute's 4 point grading scale
* Neuropathic symptoms must be related to chemotherapy (in the opinion of the treating physician)
* Patients must have had neuropathic symptoms for a minimum of 3 months
* No plans to change pain medication regimen during the course of the study
* Off active chemotherapy treatment for minimum of 3 months
* Hormonal (e.g., tamoxifen or Arimidex, etc.) and targeted (Tarceva and Avastin, etc.) therapies allowed as long as they will be continued during the course of the study
* Willing to come to one of the participating cancer centers for the therapy sessions; or willing to participate in the therapy sessions at their homes and live within a 45 minute drive of the main campuses; or can participate in the therapy sessions from MD Anderson regional care centers
* If participants agree to the Remote Training Option, participants should be willing to receive equipment at their homes and to return the equipment to MDA in case of malfunction or completion of the study
* If participants agree to the Remote Training Option, participants should be willing to download necessary software to their home computer
* If participants agree to the Remote Training Option, participants should be willing to allow research staff remote access to their computer to run the neurofeedback program

Exclusion Criteria:

* Patients who are taking any antipsychotic medications
* Patients with active central nervous system (CNS) disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy
* Patients who have ever been diagnosed with bipolar disorder or schizophrenia
* Patients with known, previously diagnosed peripheral neuropathy from causes other than chemotherapy
* Patients who have a history of head injury or who have known seizure activity
* Patients for whom any contraindications of DL are known
* Patients with suicidal ideation
* Patients who are already taking duloxetine for peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Quality Assessment Scale (PQAS) unpleasantness score | Baseline 5 up to week 10
  The primary analysis will be a linear model comparing the mean difference in the change of the unpleasantness subscale of the (PQAS)Pain Quality Assessment Scale from baseline to the end of treatment (5 weeks) between the combination arm, the duloxetine (DL), and the neurofeedback (NFB) arm while adjusting for the stratification factor. Pain Quality Assessment Scale (0-10) 0-No pain-10 Most Intense Pain Imaginable.

SECONDARY OUTCOMES:
Change in PQAS unpleasantness score | Baseline 5 up to week 10
  Will use analysis of covariance (ANCOVA) to evaluate whether chemotherapy induced peripheral neuropathy (CIPN) differs across the three subgroups with 0, 10 or 15 additional sessions of NFB, among the participants from the NFB + DL group who report at least 1-point clinical improvement in CIPN at week 5. The analysis will adjust for the baseline outcome (at week 5), time with CIPN symptoms (minimization factor), and other covariates such as age, sex, cancer stage, time since diagnosis, and cancer type, as appropriate. Pain Quality Assessment Scale (0-10) 0-No pain-10 Most Intense Pain Imaginable.
Baseline brain signatures as predictors of response to NFB and to DL | Up to week 5
  Will perform ANCOVA with the change of the unpleasantness subscale from baseline to week 5 (i.e., end of the first 15 sessions of NFB) as the outcome, intervention (NFB, DL or combo), the brain signature (one at a time) and its interaction with intervention as the independent variables of interest. Pain Quality Assessment Scale (0-10) 0-No pain-10 Most Intense Pain Imaginable.
Evaluation of patients who will require more sessions of NFB to achieve relief of symptoms | Up to 12 months post-treatment
  Linear mixed model (LMM) analyses will be performed using data measured at end of treatment, months 6 and 12 only on patients who report clinical improvement at week 5.
Change in cancer-related symptoms | Baseline up to 12 months post-treatment
  ANCOVA and LMM analyses will be performed to evaluate the effect of the number of additional NFB sessions on cancer-related symptoms.
Change in physical functioning | Baseline up to 12 months post-treatment
  ANCOVA and LMM analyses will be performed to evaluate the effect of the number of additional NFB sessions on physical functioning.
Change in quality of life | Baseline up to 12 months post-treatment
  ANCOVA and LMM analyses will be performed to evaluate the effect of the number of additional NFB sessions on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Harris Health System (LBJ), Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org